CLINICAL TRIAL: NCT04443920
Title: Comparison of the Effect of Two Common Regimens of Administration of Tranexamic Acid on Hemostasis and Clinical Outcome of Patients Undergoing Total Knee Arthroplasty
Brief Title: Tranexamic Acid for Total Knee Arthroscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1372794
Record Dates: First submitted 2020-06-15; First posted 2020-06-23 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Blood Loss, Surgical
MeSH Terms: conditions — Blood Loss, Surgical | interventions — Tranexamic Acid; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tranexamic acid (TXA) (Active Comparator): All patients will receive 15 mg/kg Tranexamic acid (TXA) IV prior to skin incision. This arm will receive a second intravenous dose of 15 mg/kg of Tranexamic acid (TXA) before the release of the tourniquet. The medication is delivered from the pharmacy in a masked syringe labeled as "study medication."
  Interventions: Drug: Tranexamic acid (TXA)
- Placebo Normal Saline (NS) (Placebo Comparator): All patients will receive 15 mg/kg Tranexamic acid (TXA) IV prior to skin incision. This arm will receive a second intravenous dose of placebo (Normal Saline) in the volume calculated to be equal to the volume of 15 mg/kg of TXA. The medication is delivered from the pharmacy in a masked syringe labeled as "study medication."
  Interventions: Drug: Placebo Normal Saline (NS)

INTERVENTIONS:
Drug: Tranexamic acid (TXA) — Randomly assigned [1:1 ratio] using a computer generated table of random numbers to 1 of the 2 intervention groups
  Other Names: Lysteda; Cyklokapron
  Arms: Tranexamic acid (TXA)
Drug: Placebo Normal Saline (NS) — Randomly assigned [1:1 ratio] using a computer generated table of random numbers to 1 of the 2 intervention groups
  Other Names: Sodium chloride
  Arms: Placebo Normal Saline (NS)

SUMMARY:
The purpose of this investigation is to determine the most effective regimen of administration of tranexamic acid to improve clinical outcome among patients undergoing total knee arthroplasty.

DETAILED DESCRIPTION:
Tranexamic acid (TXA) is synthetic lysine analog, which acts as anti-fibrinolytic agent by preventing conversion of plasminogen in to plasmin. Various regimens of TXA administration (routes, doses, timing) have been used to decrease perioperative blood loss and improve clinical outcomes among patients undergoing different orthopedic surgeries. We are conducting this prospective randomized placebo controlled trial to compare the effect of the two most common regimens of TXA administration on hemostasis and clinical outcomes among patients undergoing total knee arthroplasty. All recruited patients receive the first dose of 15mg/kg of IV TXA prior to skin incision. The second dose of 15mg/kg IV TXA or identical placebo is administered prior to the release of the tourniquet.

The assessment of hemostasis is performed using whole blood sample via viscoelastic testing by rotational thromboelastography (ROTEM). A blood sample is collected in the preoperative area and after the administration of each dose of TXA. Clinical data is collected until 90 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

- Adult patients who are scheduled to undergo total knee arthroplasty will be approached to participate.

Exclusion Criteria:

* Known allergy to TXA
* History of venous or arterial thrombosis within 12 months
* History of thromboembolic event within 12 months
* Acute ischemic event (stroke, transient ischemic attack, myocardial infarction, ischemic retinopathy) within 6 months
* Known congenital thrombophilia

Relative Contraindications:

* History of seizures
* Impaired kidney function (Glomerular filtration rate < 30 ml/min)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2019-10-29 (Actual); Primary Completion 2020-10-07 (Actual); Study Completion 2021-01-08 (Actual)

PRIMARY OUTCOMES:
Assessment of changes in hemostasis via viscoelastic testing. | intraoperative (min)
  To compare the magnitude of lysis via lysis indexes.

SECONDARY OUTCOMES:
Hematocrit | postoperative day 1
  The comparison of hematocrit recordings from preoperative period to the postoperative period
Length of Hospitalization | up to 7 days
  Length of hospital stay from day of surgery to discharge from hospital.
The number of blood transfusions | 90 days
  The number of blood products transfused after surgery
Hospital readmissions | 90 days
  The occurrence of hospital readmissions following surgery

CONTACTS AND LOCATIONS:
Overall Officials: Denis Snegovskikh, MD, Principal Investigator — Rhode Island Hospital; Brown University
Locations (1):
- Miriam Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pachauri A, Acharya KK, Tiwari AK. The effect of tranexamic acid on hemoglobin levels during total knee arthroplasty. Am J Ther. 2014 Sep-Oct;21(5):366-70. doi: 10.1097/MJT.0b013e318250f85a. PMID 23917458
- [Result] Aguilera X, Martinez-Zapata MJ, Bosch A, Urrutia G, Gonzalez JC, Jordan M, Gich I, Maymo RM, Martinez N, Monllau JC, Celaya F, Fernandez JA. Efficacy and safety of fibrin glue and tranexamic acid to prevent postoperative blood loss in total knee arthroplasty: a randomized controlled clinical trial. J Bone Joint Surg Am. 2013 Nov 20;95(22):2001-7. doi: 10.2106/JBJS.L.01182. PMID 24257657
- [Result] Kim TK, Chang CB, Kang YG, Seo ES, Lee JH, Yun JH, Lee SH. Clinical value of tranexamic acid in unilateral and simultaneous bilateral TKAs under a contemporary blood-saving protocol: a randomized controlled trial. Knee Surg Sports Traumatol Arthrosc. 2014 Aug;22(8):1870-8. doi: 10.1007/s00167-013-2492-1. Epub 2013 Apr 17. PMID 23592025
- [Result] Na HS, Shin HJ, Lee YJ, Kim JH, Koo KH, Do SH. The effect of tranexamic acid on blood coagulation in total hip replacement arthroplasty: rotational thromboelastographic (ROTEM(R)) analysis. Anaesthesia. 2016 Jan;71(1):67-75. doi: 10.1111/anae.13270. Epub 2015 Nov 12. PMID 26559015